CLINICAL TRIAL: NCT02159963
Title: High Intensity Interval Training in Patients With Facioscapulohumeral Muscular Dystrophy
Brief Title: High Intensity Training in Patients With Facioscapulohumeral Muscular Dystrophy
Acronym: HIT-FSHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grete Andersen, MD (Other)
Responsible Party: Sponsor-Investigator, Grete Andersen, MD, MD, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-4-2014-035 (FSH)
Record Dates: First submitted 2014-06-04; First posted 2014-06-10 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: FSHD - Facioscapulohumeral Muscular Dystrophy
Keywords: FSHD; HIT; Training; Exercise; 10-20-30 interval training
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supervised training (Experimental): 8 weeks of high intensity training three times a week, once supervised. Followed by 8 weeks home based, unsupervised optional training.
  Interventions: Other: Supervised training; Other: Optional training
- Unsupervised training (Experimental): Participants have 8 weeks of non-intervention "Control" period, followed by 8 weeks of home based, unsupervised high intensity interval training.
  Interventions: Other: Unsupervised training; Other: Control

INTERVENTIONS:
Other: Supervised training — 8 weeks high intensity interval training, 3 times a week, one is supervised, two are home based unsupervised.
  Arms: Supervised training
Other: Unsupervised training — 8 weeks home based high-intensity-interval cycle-training 3 times a week.
  Arms: Unsupervised training
Other: Optional training — 8 weeks of optional home based, unsupervised training.
  Arms: Supervised training
Other: Control — 8 weeks of control period. Participants are doing daily living.
  Arms: Unsupervised training

SUMMARY:
The investigators aim to investigate the effect of high-intensity training in patients with facioscapulohumeral muscular dystrophy. Can patients benefit from this type of exercise without muscle damage.

DETAILED DESCRIPTION:
Clinical trials have in recent years demonstrated that aerobic exercise, are both effective and safe in patients with facioscapulohumeral muscular dystrophy. Previous studies have tested exercise at moderate intensity. No studies have so far investigated whether high-intensity-training (HIIT) exercise can increase fitness, or the training will cause muscle damage. However, we know that patients with facioscapulohumeral muscular dystrophy do not get increased muscle damage after a single exercise at high intensity.

Investigators aim to investigate whether patients with facioscapulohumeral muscular disease may increase their fitness and improve their functioning in everyday life without muscle injury in a time-saving high intensity training.

To investigate whether HIIT is safe and effective, three groups of participants are included. Two training groups, one group of patients and another with healthy matched subjects. The training is done on an ergometer-bike three times a week for 8 weeks. One weekly training will be supervised. The training consists of an interval training program (10-20-30). The third group is a none-training control group of patients. This group will undergo the same tests as the two training groups.

To investigate wether participants would continue HIIT training after 8 weeks of supervised training, the two training groups, one group of patients and one group of healthy matched subjects, are tested after additional 8 weeks of home based optional training.

To investigate wether patients with muscular dystrophy facioscapulohumeral will perform unsupervised HIIT training and whether it will be as effective as the supervised training, the control group of patients who did not train the first 8 weeks, is instructed to do home based HIIT for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Facioscapulohumeral muscular dystrophy or
* healthy matched control, matched for age, gender, BMI and activity level.

Exclusion Criteria:

* More than 1 hour cardiac exercise weekly before inclusion.
* Pregnant or breastfeeding women.
* Physical or mental condition, which could influence the results.
* Participating in other studies, which could influence the results.
* Physical or mental condition, which prevent participating in the study protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Incremental test | week 1,6,11 and 18
  An incremental test is performed at baseline (week 1), after 4 weeks interval training, in the end of 8 weeks interval training, and after another 8 week of individual home based training. The primary outcome is change from baseline in maximal oxygen consumption and work load.

SECONDARY OUTCOMES:
Physical function | baseline, week 6,11 and 18
  We measure changes from baseline in muscle strength, walking speed and the ability to rise up from a chair.
  Muscle strength is measured by a hand-held dynamometer. Walking speed is measured by a 6 minute walk test. The ability to rise up from a chair is measured by a 5-times-sit-to-stand-test.
Self-assessment | Every day in week 1-11
  Changes between run-in period (week 1-2) and the first intervention period (week 3-11).
  Participants evaluate pain, muscle fatigue and daily activity level every day using a visual analog scale (VAS).
Creatine Kinase | week 1,6,11 and 18
  Creatine Kinase (CK) is measure in plasma at week 1,6,11 and 18 in all participants. In the supervised training participants CK is also measured once a week doing the 8 weeks of supervised training.
Activity level | baseline, week 10 and week 18.
  Change in activity level from baseline is measure as step/day. Participants is wearing a pedometer for seven days.

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen Neuromuscular Center, department of Neurology, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Andersen G, Hedermann G, Witting N, Duno M, Andersen H, Vissing J. The antimyotonic effect of lamotrigine in non-dystrophic myotonias: a double-blind randomized study. Brain. 2017 Sep 1;140(9):2295-2305. doi: 10.1093/brain/awx192. PMID 29050397
- See also: The Neuromuscular research units web-side — http://neuromuscular.dk